CLINICAL TRIAL: NCT02539277
Title: A Post-marketing Research on Jinyebaidu Granule in Treating Patients With Acute Upper Respiratory Infection: A Double Blind, Double Dummy, Randomized, Controlled Trial
Brief Title: A Post-marketing Research on Jinyebaidu Granule in Treating Patients With Acute Upper Respiratory Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: First Affiliated Hospital of Heilongjiang Chinese Medicine University (Other); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Beijing Hospital of Traditional Chinese Medicine (Other); Changchun University of Chinese Medicine (Other); Liaoning University of Traditional Chinese Medicine (Other); Shandong University of Traditional Chinese Medicine (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Junjie Jiang, assistant researcher, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20141107-3.0
Record Dates: First submitted 2015-04-18; First posted 2015-09-03 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-08

CONDITIONS: Acute Upper Respiratory Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): Jinyebaidu granule, blunt, 10g / time, three times a day; Fufangshuanghua granule placebo, blunt, 6g / time, 4 times a day.
  Interventions: Drug: Jinyebaidu granule; Drug: Fufangshuanghua granule placebo
- Control group (Active Comparator): Fufangshuanghua granule, blunt, 6g / time, 4 times a day; Jinyebaidu granule placebo, blunt, 10g / times, three times a day.
  Interventions: Drug: Fufangshuanghua granule; Drug: Jinyebaidu granule placebo

INTERVENTIONS:
Drug: Jinyebaidu granule — It is a chinese patent medicine extracted from four herbs: honeysuckle, isatis leaf, dandelion, and houttuynia cordata thunb.
  Arms: Treatment group
Drug: Fufangshuanghua granule — It is a Chinese patent medicne extracted from four herbs: honeysuckle, forsythia, radix Isatidis, andrographis paniculata.
  Arms: Control group
Drug: Jinyebaidu granule placebo — It is Jinyebaidu granule placebo.
  Arms: Control group
Drug: Fufangshuanghua granule placebo — It is Fufangshuanghua granule placebo.
  Arms: Treatment group

SUMMARY:
Study topic：A comparative effectiveness research on Jinyebaidu granule in treating patients with acute upper respiratory infection: A double blind, double dummy, randomized, controlled trial. It is a post-marketing clinical study to evaluate effectiveness, safety and cost-effectiveness on Jinyebaidu granule in treating acute upper respiratory infection.

Objectives of Study：This study aims to evaluate effectiveness, safety and cost-effectiveness on Jinyebaidu granule in treating patients with acute upper respiratory infection.

Study design：multi-center double-blind, double-dummy, randomized, controlled trial

DETAILED DESCRIPTION:
1. Inclusion criteria

   * Patients diagnosed as acute upper respiratory infection.
   * Patients with acute upper respiratory infection diagnosed as Traditional Chinese Medicine(TCM) syndrome wind-heat attacking the Lung (type of heat pathogen invading the defensive Qi of the lung).
   * Acute upper respiratory infection onset time is less than 36 hours.
   * Patients aged 18 to 70 years old.
   * Patients agreed to participate this study and sign the informed consent.
2. Effectiveness evaluation

   * TCM symptoms: fever, sore throat, cough with or without expectoration, headache, thirst, change of tongue body, tongue coating and pulse.
   * Signs: swollen tonsils, pharyngeal hyperemia.
   * Body temperature
3. Safety evaluation

   * Clinical symptoms and signs of adverse event reaction
   * Signs: blood pressure, respiration, heart rate, body temperature;
   * Routine blood test and urine routine;
   * Liver function and renal function: Alanine transaminase (ALT)、glutamic-oxalacetic transaminease(AST)、serum creatinine(SCr)、urea nitrogen(BUN) ;
   * Incidence of electrocardiogram(ECG) abnormalities.
4. Cost-effectiveness evaluation cost calculation

   * The direct medical costs include: the registration expenses, examination expenses, laboratory test expenses, Treatment costs, Chinese medicine expenses, Chinese herbal medicine expenses, western medicine expenses; Indirect medical costs: transportation costs, lost income patients; Adverse drug reactions cost: the cost of treatment due to adverse drug reactions.
   * Effect Evaluation:Symptoms and signs score, physical examination, the incidence of complications.
5. Number of participants 600 participants will be divided into two groups, the experimental group (n=300)and the control group (n=300).Each group will be stratified into three layers according to fever, sore throat, fever and sore throats. 100 patients will be included in each level.
6. Dose regimen

   * treatment group: Jinyebaidu granule, blunt, 10g/time, three times a day; Compound Shuanghua granules placebo, blunt, 6g /time, 4 times a day.
   * Control group: Compound double flowers particles, blunt, 6g/time, 4 times a day; Jinyebaidu Granule placebo, blunt, 10g/time, three times a day.
7. Course of treatment：5 days

ELIGIBILITY:
Inclusion Criteria

* Patients diagnosed as acute upper respiratory infection.
* Patients with acute upper respiratory infection diagnosed as Traditional Chinese Medicine(TCM) syndrome wind-heat attacking the Lung (type of heat pathogen invading the defensive Qi of the lung).
* Acute upper respiratory infection onset time is less than 36 hours.
* Patients aged 18 to 70 years old.
* Patients agreed to participate this study and sign the informed consent.

Exclusion Criteria:

* Patients diagnosed with suppurative tonsillitis (third degree), and chest X-ray imaging showed lung inflammation;
* White blood cell counts more than 12 E9, neutrophils more than 80%, ALT, AST, BUN, Cr more than 2 times of the normal upper limit;
* Patients with temperature lower than 37.5 degree centigrade, and without sore throat;
* Patients with temperature higher than 38.5 degree centigrade;
* Patients already receiving antibiotics or other similar drug treatment;
* Patients associated with other severe primary lung diseases, such as lung cancer, tuberculosis, pneumonia and other infectious diseases;
* Patients complicated with cardiovascular and cerebrovascular diseases, severe primary diseases of hematopoietic system, mental illness;
* Pregnant or lactating women;
* Patients with immunodeficiency resulted from organ transplantation, HIV / AIDS, or long-term use of immunosuppressive agents;
* Patients with drug allergy;
* Patients participating in other clinical trials, which influence outcome evaluation of the research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
The time to defervescence | defined as the time from the first dose of study medication to the time when the body temperature declined to lower than 37.3ºC

SECONDARY OUTCOMES:
Change of symptoms score | change from baseline symptoms score at the third day and at the fifth day
  The symptoms includes sore throat, cough, expectoration, headache, thirst. According to severity ,each symptom include four grades. The scores of sore throat are 0,2,4,6. The scores of cough, expectoration ,headache, thirst are 0,1,2,3. Compare the change from baseline all of symptoms score at the third day and at the fifth day.
  References: Mao bing, Li ting-qian, Li ming-quan, Tu jin-wen, Zhang rui-ming, et al. Clinical randomized double--blinded observation on effect of Jinyebaidu Granule in treating the disease of wind-heat attacking the lung(type of heat pathogen invading the defensive Qi of the lung). chinese JounIal of Evidence-Based Medicine Jun, 2003,3(2):115-120
Change of signs score | change from baseline signs score at the fifth day
  The signs includes swollen tonsils and pharyngeal hyperemia. According to severity, each sign includes four grades. The scores are 0,4,6,8.
  References: Mao bing, Li ting-qian, Li ming-quan, Tu jin-wen, Zhang rui-ming, et al. Clinical randomized double--blinded observation on effect of Jinyebaidu Granule in treating the disease of wind-heat attacking the lung(type of heat pathogen invading the defensive Qi of the lung). chinese JounIal of Evidence-Based Medicine Jun, 2003,3(2):115-120
Adverse events | All the time in the study
Change of routine blood test | Change from base line, on the fifth day
  The routine blood test includes white blood cell count, neutral cell ratio, lymphocyte ratio, single nuclear cell ratio, red blood cell count, hemoglobin, platelet count
Change of urine routine | Change from base line, on the fifth day
  The urine routine includes white blood cell count, red blood cell count,urine protein,urine sugar
Change of liver function | Change from base line, on the fifth day
  The liver function includes glutamic-pyruvic transaminase,glutamic-oxalacetic transaminase
Change of renal function | Change from base line, on the fifth day
  The renal function includes creatinine,usea nitrogen
Incidence of ECG abnormalities | Change from base line, on the fifth day

CONTACTS AND LOCATIONS:
Overall Officials: Yanming Xie, Study Chair — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, Beijing, Beijing Municipality, China